CLINICAL TRIAL: NCT03930550
Title: Infrared Transillumination of the Front of the Neck as an Aid for Awake Intubation
Brief Title: Infrared Transillumination of the Front of the Neck
Acronym: IRRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Seltz Kristensen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-18038322 IRRIS
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Tracheal Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infrared guidance first (Experimental): In this arm the infra red guidance is applied to the first passage of the flexible scope to the trachea.
  The second passage of the flexible scope is without the infrared light
  Interventions: Procedure: Tracheal intubation by endoscopy with flexible bronchoscope
- Infrared guidance last (Active Comparator): In this arm NO infra red guidance is applied to the first passage of the flexible scope to the trachea.
  The second passage of the flexible scope is with the infrared light as guide
  Interventions: Procedure: Tracheal intubation by endoscopy with flexible bronchoscope

INTERVENTIONS:
Procedure: Tracheal intubation by endoscopy with flexible bronchoscope — A blinking infrared light source is placed on the anterior neck at the level of the cricothyroid membrane to serve as a guide to facilitate finding the way to the trachea

SUMMARY:
Infrared light is applied to the front of the neck of patients for awake flexible optical intubation. The infrared light can be detected by the camera at the tip of the flexible video-bronchoscope. The flexible scope is introduced into the trachea with or without the aid of the blinking infra red light and the ease of placement of the flexible scope is studied.

DETAILED DESCRIPTION:
The investigators study patients for anaesthesia who will need endotracheal intubation and in whom the intubation is predicted to become difficult so that an awake flexible-video-scope-guided intubation is chosen.

Infrared light is applied to the front of the neck of patients for awake flexible optical intubation. The infrared light can be detected by the camera at the tip of the flexible video-bronchoscope. The flexible scope is introduced into the trachea with or without the aid of the blinking infra red light and the ease of placement of the flexible scope is studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for awake tracheal intubation over the insertion cord of a flexible video-trachea-bronchoscope.

Exclusion Criteria:

* Age < 18 years
* Patients at high risk of aspiration of gastric content
* Patients with hypoxia, saturation < 90 % on ambient air
* Patients with audible stridor at rest
* American Society of Anesthesiology (ASA) physical class > 3
* contraindication for trans-crico-thyoid-membrane puncture (cancer, infection on the site, severely coagulopathies, inability to identify the crico-thyroid membrane)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Fraction of cases where the blinking light is seen before the vocal cords are seen | 1 day of the procedure
  The flexible scope is entered into the airway twice, . It is noted from watching the videos of the procedures if the blinking light or the vocal cords are seen first -

SECONDARY OUTCOMES:
Fraction of cases where the blinking light is seen from the teeth, the mouth, the pharynx and the larynx and the fra fraction of cases where the vocal cords are seen from the teeth, the mouth, the pharynx and the larynx | 1 day of the procedure
  The flexible scope is entered into the airway twice, one time with and one time without the blinking light on the front of the neck. It is noted from watching the videos of the procedures if the blinking light or the vocal cords are seen first - and from which anatomical location it is seen.
Time from the tip of the flexible scope passes the teeth until vocal cords are seen | 1 day of the procedure
  Time measured from the tip of the flexible scope passes the teeth until the vocal cords are seen

OTHER OUTCOMES:
Time from the tip of the flexible scope passes the teeth until the blinking light is seen | 1 day of the procedure
  Time measured from the tip of the flexible scope passes the teeth until the blinking light is seen
Time from the tip of the flexible scope passes the teeth until it is at the level of the mid trachea, trachea rings are seen | 1 day of the procedure
  Time measured from the tip of the flexible scope passes the teeth until it is at the level of the mid trachea, trachea rings are seen
Number of times that the flexible scope is pulled backwards | 1 day of the procedure
  Counting the number of times that the flexible scope is pulled backwards
Number of times that the flexible scope is reinserted past the teeth | 1 day of the procedure
  Counting the number of times that the flexible scope is reinserted past the teeth
Number of times that the flexible scope touches the mucosa until the tip is in the mid-trachea | 1 day of the procedure
  Counting the Number of times that the flexible scope touches the mucosa until the tip is in the mid-trachea
Time from the flexible scope passes the teeth until a carbon dioxide (CO2) curve is seen | 1 day of the procedure
  Measuring the time from the flexible scope passes the teeth until a CO2 curve is seen on the capnograph
Oxygen saturation | 1 day of the procedure
  Oxygen saturation measured with pulse oximetry without added oxygen, with nasal oxygen, and the lowest value measured during the whole procedure.
The operators evaluation of the ease of seeing the entrance to the trachea (at the level of the vocal cords) | 1 day of the procedure
  The operators evaluation of the ease of seeing the entrance to the trachea (at the level of the vocal cords), measured on a scale from 1-10, 1=impossible, 10= very easy)
If the operator means that the blinking infra-red guidance is beneficial for the procedure, | 1 day of the procedure
  If the operator means that the blinking infra-red guidance is beneficial for the procedure, from 1 to 10, where 1= Not beneficial, 10 = extremely beneficial
If the operator can distinguish the light from trachea fro the surrounding structures? | 1 day of the procedure
  If the operator can distinguish the light from trachea fro the surrounding structures? On a scale from 1 to 10, 1= Not distinguishable, 10 = Clearly distinguishable
Operators evaluation about the ease of using the blinking light as a guide for insertion of the insertion cord of the flexible scope | 1 day of the procedure
  Operators evaluation about the ease of using the blinking light as a guide for insertion of the insertion cord of the flexible scope. On a scale from 1-10, 1= Very difficult, 10 = very easy
Fraction pf cases where there is redness of the skin on the anterior neck | 1 day of the procedure
  Observation of the skin on the anterior neck immediately after removal of the light-source, and one hour after arrival in the post-operative-recovery unit.
Time for ultrasound-guided identification of the cricothyroid membrane and for cannula cricothyroidotomy | 1 day of the procedure
  Time for ultrasound-guided identification of the cricothyroid membrane and for cannula cricothyroidotomy, measured on video of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Kristensen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, section for anaesthesia for ENT and Maxillofacial surgery, section 3071, Copenhagen, Denmark

REFERENCES:
- [Derived] Kristensen MS, Hesselfeldt R, Brinkenfeldt HK, Biro P. Infrared flashing light through the cricothyroid membrane as guidance to awake intubation with a flexible bronchoscope: A randomised cross-over study. Acta Anaesthesiol Scand. 2023 Apr;67(4):432-439. doi: 10.1111/aas.14204. Epub 2023 Feb 2. PMID 36690598